CLINICAL TRIAL: NCT05722977
Title: Surufatinib Combined With Envafolimab Followed by Surufatinib as Second or More - Line Therapy for Advanced Soft Tissue Sarcoma in a Single-arm, Phase II Study
Brief Title: Surufatinib and Envafolimab as Second or More-line Therapy in Advanced Soft Tissue Sarcoma Patients
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, WangXiang, chief physician, Peking Union Medical College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Slufenvo
Record Dates: First submitted 2023-02-01; First posted 2023-02-10 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Efficacy and Safety of Surufatinib Combined With Envafolimab as Second or More-line Therapy in Advanced Soft Tissue Sarcoma Patients
MeSH Terms: interventions — surufatinib; envafolimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Surufatinib+envafolimab (Experimental)
  Interventions: Drug: Surufatinib + envafolimab

INTERVENTIONS:
Drug: Surufatinib + envafolimab — Surufatinib: oral, fix dose 250mg, once a day; Envafolimab: subcutaneous injection, fix dose 300mg, once every three weeks

SUMMARY:
In this study, we investigated the efficacy and safty of surufatinib combined with envafolimab followed by surufatinib as second or more - line therapy in advanced soft tissue sarcoma patients. Patients who have failed at least the first-line therapy and have progressive disease or cannot tolerate within 6 months before enrollment will be treated with surufatinib combined with envafolimab.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged from 18 to 75 years old;
2. Subjects with histologically confirmed unresectable locally advanced or metastatic soft tissue sarcoma, which includes synoviosarcoma, leiomyosarcoma, undifferentiated pleomorphic sarcoma/malignant fibrous histiocytoma, fibrosarcoma, epithelioid sarcoma, angiosarcoma, alveolar soft-part sarcoma, etc. Chondrosarcoma, osteosarcoma, dermatofibrosarcoma protuberans, gastrointestinal stromal tumor and malignant mesothelioma are excluded;
3. Patients who have at least failed first-line treatment and had a disease progression within 6 months or can not tolerate the treatment. Notes: if the cumulative dose of anthracycline drugs reach threshold according to the guideline of Chinese Society of Clinical Oncology(CSCO) published in 2020, it will be regarded as intolerable;
4. Disease must be measurable by Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1). Previously irradiated focus can be considered as measurable only if there is definite progress after radiotherapy;
5. Newly obtained or archived tumor tissue samples can be provided;
6. Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 to 2 at trial entry;
7. Estimated life expectancy of more than 12 weeks;
8. Adequate organ functions defined by the protocol;
9. Negative blood pregnancy test at Screening for women of childbearing potential within 1 week before the first medication; Highly effective contraception for both male and female subjects if the risk of conception exists;
10. Able to comply with the research protocol and follow-up process for treatment and follow-up;
11. Already signed an informed consent form

Exclusion Criteria:

1. Patients whose tumors are judged by the investigators to be at high risk of invading vital blood vessels and causing fatal hemorrhage during the study.
2. Occurrence of arterial/venous thrombotic events within 6 months before treatment, such as cerebrovascular accident (including transient ischemic attack, hematencephalon and cerebral infarction), deep vein thrombosis , pulmonary embolism, etc.
3. Occurrence of clinically significant hemoptysis(>5ml fresh blood in 4 weeks), hemorrhagic tendency(bleeding>30ml within 3 months), such as gastrointestinal bleeding, hemorrhagic gastric ulcer, fecal occult blood test(FOBT) ++ in the baseline period , or vasculitis, etc;
4. Hypertension that cannot be controlled stably by drugs, which is defined as: systolic blood pressure>140mmHg or diastolic blood pressure>90mmHg;
5. With clinically significant cardiovascular diseases, including but not limited to: acute myocardial infarction, severe/unstable angina pectoris or coronary artery bypass grafting within 6 months before enrollment; congestive heart failure with New York Heart Association (NYHA) grade≥2; cardiac revascularization, hemodynamic unstable arrhythmia; Left ventricular ejection fraction(LVEF) <50%
6. QTc interval ≥ 480 milliseconds (ms) on electrocardiogram (ECG);
7. 24-h urinary protein level >1.0g/day;
8. Serum potassium, calcium (after correction for ionic or albumin-bound type) or magnesium are beyond the normal range and have clinical significance.
9. Abnormal coagulation function (INR>1.5 or PT>ULN+4s or APTT >1.5 ULN), hemorrhagic tendency or being treated with thrombolysis or anticoagulation therapy. Notes: on the premise of INR ≤ 1.5, it is allowed to use low-dose heparin (daily dosage of adults is 6000-12000U) or low-dose aspirin (daily dosage ≤ 100mg) for preventive purposes;
10. With factors affecting oral drug administration: dysphagia, post-gastrointestinal resection, chronic diarrhea and intestinal obstruction, etc
11. Presence of known active central nervous system metastasis and/or cancerous meningitis;
12. With any active, known or suspected autoimmune disease (subjects who are in stable status and do not need systemic immunosuppressant are allowed to be enrolled, such as subjects with type 1 diabetes, hypothyroidism requiring hormone replacement therapy only, skin diseases (leucoderma, psoriasis or alopecia) without the need for systemic treatment or subjects whose situation is not expected to reappear without extrinsic incentive);
13. Patients who are receiving systemic steroid treatment within 3 days before the first dose of trial drugs or any other form of immunosuppressive drugs. Notes: a. Corticosteroids can be used to deal with adverse reactions (AEs) and serious adverse reactions (SAEs) after period 1, and can also be used as a pre-medication for the control chemotherapy group, as a preventive drug for the allergy/reaction of intravenous contrast enhanced radiography, or if it is considered necessary for the subject to use. b. Except for the subjects who are receiving steroid replacement therapy every day. A daily dose of 5-7.5 mg of prednisone is an alternative treatment. c. Equivalent dose of hydrocortisone treatment can also be allowed to enter the trial if it is an alternative treatment.
14. With any clinically significant active infection, including but not limited to: active tuberculosis, infection of Human immunodeficiency virus (HIV);
15. HBV DNA of patients with chronic hepatitis B virus (HBV) infection must be <100 IU/mL, and antiviral treatment should be carried out at the same time;
16. Previous malignant disease within the last 5 years with the exception of post radical resection of basal or squamous cell carcinoma of the skin or cervical carcinoma in situ;
17. Anticancer treatment within 4 weeks before the research, including but not limited to: chemotherapy, radical radiotherapy, targeted therapy, immunotherapy, antitumor traditional Chinese medicine/ Chinese patent medicine, transcatheter arterial chemoembolization, Cryoablation or radiofrequency ablation of liver metastases;
18. History of receiving anti-angiogenic drugs such as surufatinib, bevacizumab, ramucirumab, aflibercept, anlotinib, apatinib, lenvatinib, sorafenib, sunitinib, regorafenib, fruquintinib, endostatin, etc.
19. History of receiving anti-PD-1, anti-PD-L1 or anti-PD-L2 drugs or drugs directly acting on another stimulatory or co-inhibitory T cell receptor (such as CTLA-4, OX-40, CD137, LAG3);
20. History of allergy to any component of surufatinib and envafolimab;
21. Accination with live or live/attenuated viruses within 4 weeks of the first dose of surufatinib/ envafolimab and while on trial is prohibited;
22. Have major surgery, severe traumatic injuries, fracture or ulcer within 4 weeks before treatment;
23. Pregnant or lactating women;
24. Participate in other clinical trials at present or within four weeks before enrollment;
25. According to the judgment of the researchers, the subject has other factors that may lead to the forced termination of the study, such as other severe diseases (including mental diseases) which need to be treated together, severe laboratory abnormalities , family or social factors.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-02-02 (Estimated); Primary Completion 2026-02-02 (Estimated); Study Completion 2027-02-02 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | It will be evaluated at about 18 weeks
  Assess ORR, defined as Investigator-assessed CR+PR, per RECIST 1.1.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | From the start of randomization to a minimum of 42 months
  PFS is defined as time (in months) from date of randomization to the date of the first documentation of objective progressive disease (PD) or death due to any cause in the absence of documented PD (whichever occurs first). PFS will be determined according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) based on investigator response assessment.
Disease Control Rate (DCR) | From the start of randomization to a minimum of 42 months
  Percentage of patients with CR/PR/SD in the number of patients that whose tumour can be evaluated.
Overall Survival (OS) | From the start of randomization to a minimum of 42 months
  OS is defined as the time (in months) from randomization to the date of death, regardless of the actual cause of the subject's death.
Number of Subjects With Treatment-Emergent Adverse Events (TEAEs) According to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5.0 | From the start of randomization to a minimum of 42 months
  TEAEs will be defined as the adverse events (AEs) that occur between first dose of study drug administration and 28 days after the last dose of study drug administration that were absent before treatment or that worsened relative to pretreatment state.